CLINICAL TRIAL: NCT06701448
Title: Comparative Performance of Robotic, Electromagnetic Navigation and Fluoroscopy Drives Optimal Diagnostic Strategy for Peripheral Pulmonary Lesions: a Prospective, Multi-center, Parallel-Controlled Trial
Brief Title: Comparative Performance of Robotic, Electromagnetic Navigation and Fluoroscopy Drives Optimal Diagnostic Strategy for Peripheral Pulmonary Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professor, Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EC-2022-037 (QX)-02
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Nodule; Bronchoscopy
Keywords: peripheral pulmonary lesions; optimal strategy; robotic bronchocospy; electromagnetic navigation bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RBS group (Other): Biopsy of peripheral pulmonary lesions using RBS
  Interventions: Diagnostic Test: robotic bronchosopy
- ENB group (Other): Biopsy of peripheral pulmonary lesions using ENB
  Interventions: Diagnostic Test: Electromagnetic Navigation Bronchoscopy
- FB group (Other): Biopsy of peripheral pulmonary lesions using FB
  Interventions: Diagnostic Test: Fluoroscopy bronchoscopy

INTERVENTIONS:
Diagnostic Test: robotic bronchosopy — robotic bronchoscopy
  Arms: RBS group
Diagnostic Test: Electromagnetic Navigation Bronchoscopy — Electromagnetic Navigation Bronchoscopy
  Arms: ENB group
Diagnostic Test: Fluoroscopy bronchoscopy — Fluoroscopy bronchoscopy
  Arms: FB group

SUMMARY:
Currently, the optimal method for Peripheral Pulmonary Lesions (PPL) is uncertain. We aim to compare the diagnostic yield of Robotic Bronchoscopy System (RBS), Electromagnetic Navigation Bronchoscopy (ENB), Fluoroscope-Bronchoscopy (FB).

DETAILED DESCRIPTION:
Pulmonary peripheral lesions (PPLs) are a prevalent medical condition and a significant contributory factor to the widespread health and social issues associated with pulmonary diseases, particularly lung cancer. In China, lung cancer has become the most common cancer in terms of new cases and deaths, with 1,060,600 new cases and 736,600 deaths recorded. Early diagnosis of PPLs is essential to prevent their progression to cancer.

Fluoroscopy bronchoscopy (FB) was previously the primary diagnostic method for PPLs. However, its limitation lies in the occurrence of adverse events, particularly pneumothorax. Furthermore, many patients are not suitable for percutaneous biopsy which has led to the exploration of alternative methods for diagnosis.

With the advancement of bronchoscopy, several innovative technologies have been proposed and developed for sampling tissues from PPLs in recent years. Electromagnetic navigation bronchoscopy (ENB) stands out as one of the most superior among them. Its integration of real-time guidance and precise maneuverability of a biopsy instrument gives it an advantage over alternative technologies.

The Robotic Bronchoscopy System (RBS) offers an excellent alternative method with enhanced flexibility and stability. The bronchoscopist is able to control the insertion and biopsy of the RBS from a console located near the patient, allowing for a more stable posture to access the distal airway compared to conventional bronchoscopy. Numerous studies have demonstrated that RBS exhibits an excellent navigation success rate and diagnosis rate. A multi-center study on the ION endoluminal platform (Intuitive Surgical, Inc.) revealed a navigation yield as high as 98.7% and a total diagnostic yield of 81.7%. Similarly, research on the Monarch RAB showed navigation yield and diagnostic yield of 96.2% and 74.1%, respectively.

The iLung Infinity system (LungHealth MedTech Ltd, Shanghai, China) is specifically designed to utilize real-time electromagnetic technology in order to localize and guide bronchoscopic tools towards the lesion on a pre-constructed three-dimensional bronchial tree.

The Unicorn Kylin™ robotic system represents a novel Robotic Bronchoscopy System (RBS). The system comprises an unit with two mechanical arms boasting nine degrees of freedom, a flexible bronchoscope (outer diameter: 4.3 mm; Working channel: 2.0 mm), and a console equipped with electromagnetic navigation system.

In the clinical setting, different sampling methods have a crucial impact on the quality of tissue samples and the treatment of patients. However, there are currently no existing studies that directly compare the diagnostic performance of RBS, ENB, and FB using the same definition of diagnostic yield in a homogenous patient population. It is imperative to gather comparative effectiveness data on these systems in order to develop an optimal strategy for patient care. Therefore, this study aimed to assess the diagnostic performance of RBS, ENB, and FB when conducting peripheral pulmonary biopsies. To achieve this goal, a multicenter controlled study was conducted across six medical centers or hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion if they meet all of the following criteria:

  1. Age ≥18 years and ≤75 years, with no gender restrictions;
  2. Presence of a peripheral lung lesion on chest CT
  3. Patients voluntarily agree to undergo bronchoscopy and meet the requirements for the procedure;
  4. patients are capable of understanding the purpose of the trial, demonstrate good compliance with the examinations and follow-up, voluntarily participate in the clinical trial, and sign an informed consent form.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from this study:

  1. Presence of contraindications for bronchoscopy, including: active massive hemoptysis; recent myocardial infarction or unstable angina; severe cardiac or pulmonary dysfunction; severe hypertension and arrhythmias; uncorrectable bleeding tendencies or severe coagulation disorders (such as platelet count <60×10^9/L), uremia; severe pulmonary artery hypertension; severe superior vena cava syndrome; intracranial hypertension; acute cerebrovascular events; aortic dissection or aneurysm; multiple bullae; extreme systemic exhaustion;
  2. Female patients who are breastfeeding, pregnant, or planning pregnancy;
  3. Patients with electromagnetic active implantable medical devices;
  4. Subjects allergic to anesthetics; or with a history of multiple severe allergies, hereditary allergy history;
  5. Those who have participated in or are currently participating in drug clinical trials within 3 months before screening, or have participated in other medical device clinical trials within 30 days;
  6. Any other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall diagnostic yield | 1 years after biopsy
  Overall diagnostic yield was considered as the primary outcome, defined as the number of cases in which the diagnosis of bronchoscopy matched the final diagnosis, divided by the total number of completed cases during follow-up. A lesion was considered malignant if tumor cells were found in histological and/or cytological specimens. It was considered benign if pathological evaluation showed specific benign pathology and/or non-specific benign lesions confirmed by MDT discussion.

SECONDARY OUTCOMES:
Strict diagnostic yield | 7 days after biopsy
  The secondary outcome of interest was the strict diagnostic yield, which is defined as the proportion of cases diagnosed with bronchoscopy pathology divided by all cases sampled using a specific technology. The bronchoscopy pathology diagnosis only included malignant and specific benign lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong 510163, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skouras VS, Gkiozos I, Charpidou AG, Syrigos KN. Robotic Bronchoscopy in Lung Cancer Diagnosis. Cancers (Basel). 2024 Mar 17;16(6):1179. doi: 10.3390/cancers16061179. PMID 38539514